CLINICAL TRIAL: NCT00627263
Title: Reducing Vulnerability to ICD Shock Treated Ventricular Arrhythmias
Brief Title: Stress Reduction to Reduce Risk for Arrhythmia in ICD Patients (The RISTA Study)
Acronym: RISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0708003000; R01HL084438 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Arrhythmias, Cardiac
Keywords: ICD; Cardiac Arrhythmia; Arrhythmia; Stress; Anger
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Participants will receive the usual cardiologic care for ICD patients provided by their medical team.
- 2 (Experimental): In addition to the usual cardiologic care for ICD patients provided by the participants medical team, those randomized to Intervention will receive the stress reduction treatment (SRT) program (see below).
  Interventions: Behavioral: Stress reduction treatment (SRT) program

INTERVENTIONS:
Behavioral: Stress reduction treatment (SRT) program — The SRT program is a cognitive behavioral program that consists of 8 group sessions over a period of 10 weeks.
  Arms: 2

SUMMARY:
An implantable cardioverter defibrillator (ICD) is a small device that is implanted in the chest and uses electrical shocks to control arrhythmias, which are abnormal heart rhythms. Arrhythmias can be caused by many factors, including stress and anger. This study will evaluate the use of a stress reduction treatment (SRT) program aimed at reducing the occurrence of arrhythmias that require treatment with an ICD shock.

DETAILED DESCRIPTION:
An ICD is a device designed to quickly detect a life-threatening, rapid heartbeat. Through a process called defibrillation, the ICD tries to convert an abnormal heart rhythm back to normal by delivering an electrical shock to the heart. The ICD continuously monitors heartbeats to ensure that they are normal, and it only delivers a shock to the heart when it senses a life-threatening arrhythmia. Because of the recent funding approval by Medicaid, it is now estimated that more than 500,000 people will receive ICDs annually. Although ICDs are life-saving medical devices, some people may experience anxiety, depression, and impaired quality of life as a result of the repeated ICD shocks. Additionally, increased mental and emotional stress and anger may increase the likelihood of experiencing more arrhythmias requiring an ICD shock. SRT programs that encourage people to manage their emotions may decrease the frequency of arrhythmias. Furthermore, SRT programs have been shown to be successful at reducing other stress-related heart conditions. The purpose of this study is to evaluate the effectiveness of an SRT program at reducing the incidence of ICD shock-treated arrhythmias among people with newly implanted ICDs.

This study will enroll people who have recently received an ICD. Initially, participants will complete questionnaires about mood and attitudes. Next, at a baseline study visit, participants will complete a mental stress exercise in which they will perform math problems and describe an experience that made them angry. During this exercise, participants will undergo blood pressure measurements, blood collection, and an electrocardiogram (EKG) to measure electrical activity of the heart. Participants will also wear a monitor for 24 hours after the study visit to record heart activity. Participants will then be randomly assigned to either take part in the SRT group and receive usual care or only receive usual care. For 10 weeks, participants in the SRT group will attend 8 group sessions that will focus on learning and applying stress reduction techniques to everyday living. All participants will attend a 3-month follow-up visit for repeat baseline testing. At Months 6, 12, and 24, participants will complete questionnaires during routine doctor's visits or by mail.

ELIGIBILITY:
Inclusion Criteria:

* Receiving an ICD or currently have an ICD and have recieved appropriated ICD shock therapy in the 6 months before study entry
* Ischemic cardiomyopathy or non-ischemic (dilated) cardiomyopathy
* Fluent in spoken and written English
* Able to participate in the SRT program

Exclusion Criteria:

* Unable to comply with the study or participate in SRT treatment, if assigned
* Incapacitating illness (e.g., stage IV congestive heart failure) that would interfere with study participation
* Life expectancy of less than 2 years (e.g., due to metastatic cancer)
* Uncommon etiologies of arrhythmia (e.g., long QT syndrome, hypertrophic cardiomyopathy, Brugada syndrome)
* Cognitive impairment, based on Mini-Mental Status Exam (MMSE) and educational level. If education level is less than 8th grade, then people with an MMSE score of less than 17 will not be enrolled; if education level is greater than 8th grade, then people with an MMSE score of less than 24 will not be enrolled.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ICD shock-treated ventricular arrhythmia event-free survival | Measured at Month 24
  The occurrence of ICD shock treated ventricular arrhythmia

SECONDARY OUTCOMES:
Laboratory stress-provoked arrhythmogenic changes in the heart rhythm | Measured at Baseline and Month 6
  Arrhythmogenic changes in the heart rhythm during laboratory mental stress
24-hour heart rate variability | Measured at Baseline and Month 6
  Heart rate variability on 24 hour holter monitoring
Quality of life | Measured at Month 24
  SF-36 assessment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Burg, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University Medical School, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Donahue RG, Lampert R, Dornelas E, Clemow L, Burg MM; RISTA Investigators. Rationale and design of a randomized clinical trial comparing stress reduction treatment to usual cardiac care: the Reducing Vulnerability to Implantable Cardioverter Defibrillator Shock-Treated Ventricular Arrhythmias (RISTA) trial. Psychosom Med. 2010 Feb;72(2):172-7. doi: 10.1097/PSY.0b013e3181c932d4. Epub 2009 Dec 22. PMID 20028832